CLINICAL TRIAL: NCT03553693
Title: Optimizing HIV Viral Load Monitoring and Outcomes for High Risk Populations
Brief Title: Rapid HIV Viral Load Monitoring in High Risk Patients In Uganda
Acronym: RAPID-VL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RAPID-VL
Record Dates: First submitted 2018-05-18; First posted 2018-06-12 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-01

CONDITIONS: HIV
Keywords: HIV; Viral Load; Counseling; Costs and Costs Analysis; Point-Of-Care Systems

STUDY DESIGN:
Intervention Model Description: Comparative effectiveness cluster-randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Clinics (Experimental): RAPID-VL study intervention testing and counseling package, which includes near point-of-care viral load (VL) testing at local testing hubs, structured VL counseling, forms to track VL ordering and testing, with feedback and performance evaluations at regular intervals.
  Interventions: Other: RAPID-VL study intervention
- Control Clinics (No Intervention): Standard of care VL testing and counseling procedures consistent with country guidelines.

INTERVENTIONS:
Other: RAPID-VL study intervention — * Viral load (VL) ordering flowsheet with periodic health facility performance feedback
  * Rapid near-point-of-care VL testing and telephone delivery of results
  * Structured VL counseling package
  Arms: Intervention Clinics

SUMMARY:
The RAPID-VL study will take place in 20 HIV care health facilities in Southwestern Uganda. The study will test the hypothesis that a multi-component intervention package that targets barriers to efficient and timely HIV viral load (VL) testing will improve test ordering, speed up result turnaround times, and improve the quality of VL results counseling to patients. Phase 1 of the study will consist of a 1-year retrospective medical record review in all participating health facilities. In Phase 2 the intervention will be introduced in 10 randomly chosen health facilities, while the remaining 10 sites will continue with standard VL testing and counseling operations. The study will measure the speed and efficiency of VL testing, experiences of patients and clinicians with the intervention, and the cost of the intervention.

DETAILED DESCRIPTION:
We will test the hypothesis that a multi-component intervention grounded in implementation science principles and that targets key barriers to optimal HIV viral load (VL) processing will improve viral load ordering, speed up viral load turnaround, and improve the quality of viral load counseling of results to patients within a Ugandan network of HIV care clinics. Specific objectives are as follows: Objective 1: Determine the comparative effectiveness of the RAPID-VL intervention on VL ordering and VL turnaround time: We will randomize 20 HIV clinics to the RAPID-VL multi-component intervention vs. standard of care VL procedures (n=10 clinics each, 60 patients/health facility). Objective 2: Identify facilitators and barriers to implementation, and perceived utility of the RAPID-VL intervention from both the patient and clinician perspectives. Objective 3: Determine the costs, cost-effectiveness, and incremental change costs of the RAPID-VL intervention.

ELIGIBILITY:
Inclusion Criteria:

Phase 1, Intervention and Control Clinics:

"High risk" subgroups of patients (n=10 each per clinic, total of 40 per clinic): registered for care, with a clinic visit within a year of the Phase 1 start date, plus the following:

1. Pregnant or breastfeeding women: Inclusion criteria: (1) pregnant or breastfeeding at any time during Phase 1, confirmed by clinic documentation
2. Children/adolescents: Inclusion criteria: (1) age 2-17 years, (2) no documentation of pregnancy in clinical record
3. Persons with most recent VL unsuppressed (i.e. detectable): Inclusion criteria: (1) any age, (2) most recent VL documented in the medical record within the last 1 year, with a value of >1000 copies/mL on any assay, (3) no documentation of pregnancy in clinical record
4. Persons with no VL in last one year: Inclusion criteria: (1) any age, (2) last VL is dated >1 year ago (if ever started on ART) or no VL on file (if never started ART) (3) no documentation of pregnancy in clinical record

"Non-high-risk" patients (n=20 per clinic): Inclusion criteria (1) adult (age ≥18 years), (2) registered for care, with clinic visit within a year of the Phase 1 start date, (3) already on ART or starting ART at time of study enrollment, (4) do not meet any of the inclusion criteria of a "high risk" subgroup

Phase 2, Intervention Clinics:

We will select 60 patients in each of the 10 intervention clinics (600 patients total; different than the 60 patients in each clinic studied in Phase 1), with inclusion criteria as follows:

"High risk" subgroups of patients (n=10 each per clinic, total of 40 per clinic): registered for care, with a clinic visit within a year of the Phase 2 start date; able to consent for study participation; plus the following:

1. Pregnant or breastfeeding women: Inclusion criteria: (1) currently pregnant or breastfeeding, confirmed by clinic standard documentation
2. Children/adolescents: Inclusion criteria: (1) age 2-17 years, (2) parent/guardian able and willing to provide affirmative consent for study participation, except in the case of mature or emancipated minors, (3) no documentation of pregnancy in the clinic record
3. Persons with most recent VL unsuppressed: Inclusion criteria: (1) any age, (2) most recent VL documented in the medical record within the last 1 year, with a value of >1000 copies/mL on any assay, (3) no documentation of pregnancy in the clinical record
4. Persons with no VL in last 1 year: Inclusion criteria: (1) any age, (2) last VL is dated >1 year ago (if ever started ART) or no VL on file (if never started ART , (3) no documentation of pregnancy in the clinical record

"Non-high-risk" patients (n=20 per clinic): Inclusion criteria: (1) adult (age ≥18 years), (2) registered in the general HIV clinic, (3) already on ART or starting ART at time of study enrollment, (4) do not meet any of the inclusion criteria of a "high risk" subgroup

Phase 2, Control Clinics:

We will select 60 patients in each of the 10 control clinics (600 patients total; different than the 60 patients in each clinic studied in Phase 1), with inclusion criteria as follows

"High risk" subgroups of patients (n=10 each per clinic, total of 40 per clinic): registered for care, with a clinic visit within a year of the Phase 1 start date; able to provide consent; plus the following:

1. Pregnant or breastfeeding women: Inclusion criteria: (1) pregnant or breastfeeding at any time during Phase 2, confirmed by clinic documentation
2. Children/adolescents: Inclusion criteria: (1) age 2-17 years, (2) parent/guardian able and willing to provide affirmative consent for study participation, except in the case of mature or emancipated minors, (3) no documentation of pregnancy in clinical record
3. Persons with most recent VL suppressed: Inclusion criteria: (1) any age, (2) most recent VL documented in the medical record within the last 1 year, with a value of >1000 copies/mL on any assay, (3) no documentation of pregnancy in clinical record
4. Persons with no VL in last 1 year: Inclusion criteria: (1) any age, (2) last VL is dated >1 year ago (if ever started ART) or no VL on file (if never started ART), (3) no documentation of pregnancy in clinical record

"Non-high-risk" patients (n=20 per clinic): Inclusion criteria: (1) adult (age ≥18 years), (2) registered for care, with clinic visit within a year of the Phase 2 start date, (3) already on ART or starting ART at time of study enrollment, (4) do not meet any of the inclusion criteria of a "high risk" subgroup

Exclusion criteria: None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2443 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

PRIMARY OUTCOMES:
Successful VL ordering | 1 year
  Proportion of patients who had a VL ordered when indicated by country guidelines
VL turnaround time | 1 year
  Mean turnaround time in days from VL ordering to delivery of results to patient

SECONDARY OUTCOMES:
VL suppression 12 months after the start of Phase 2 of trial | 12 months after the start of Phase 2 of trial
  Proportion of subjects suppressed 12 months after start of RAPID-VL participation
Viral re-suppression after positive VL | 1 year
  Proportion of patients with a positive (unsuppressed) VL whose next subsequent VL was suppressed
Number of patients changed from 1st line to 2nd line ART | 1 year
  Number of patients who switched to a 2nd line ART regimen for any reason
CPHL integration process | 12 months after the start of Phase 2 of trial
  Establishment of a process for data transfer to Uganda's Central Public Health Laboratory (CPHL) (yes/no)
VL results in CPHL database | 12 months after the start of Phase 2 of trial
  Proportion of VL results generated in study that are present in CPHL database at study end

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Jain, MD, MAS, Principal Investigator — University of California, San Francisco; Moses R Kamya, MBChB, MMed, Principal Investigator — Makerere University
Locations (1):
- Southwestern Uganda, Mbarara, Uganda

REFERENCES:
- [Background] Working Group on Modelling of Antiretroviral Therapy Monitoring Strategies in Sub-Saharan Africa; Phillips A, Shroufi A, Vojnov L, Cohn J, Roberts T, Ellman T, Bonner K, Rousseau C, Garnett G, Cambiano V, Nakagawa F, Ford D, Bansi-Matharu L, Miners A, Lundgren JD, Eaton JW, Parkes-Ratanshi R, Katz Z, Maman D, Ford N, Vitoria M, Doherty M, Dowdy D, Nichols B, Murtagh M, Wareham M, Palamountain KM, Chakanyuka Musanhu C, Stevens W, Katzenstein D, Ciaranello A, Barnabas R, Braithwaite RS, Bendavid E, Nathoo KJ, van de Vijver D, Wilson DP, Holmes C, Bershteyn A, Walker S, Raizes E, Jani I, Nelson LJ, Peeling R, Terris-Prestholt F, Murungu J, Mutasa-Apollo T, Hallett TB, Revill P. Sustainable HIV treatment in Africa through viral-load-informed differentiated care. Nature. 2015 Dec 3;528(7580):S68-76. doi: 10.1038/nature16046. PMID 26633768
- [Background] Rutstein SE, Golin CE, Wheeler SB, Kamwendo D, Hosseinipour MC, Weinberger M, Miller WC, Biddle AK, Soko A, Mkandawire M, Mwenda R, Sarr A, Gupta S, Mataya R. On the front line of HIV virological monitoring: barriers and facilitators from a provider perspective in resource-limited settings. AIDS Care. 2016;28(1):1-10. doi: 10.1080/09540121.2015.1058896. Epub 2015 Aug 17. PMID 26278724
- [Background] Roberts T, Cohn J, Bonner K, Hargreaves S. Scale-up of Routine Viral Load Testing in Resource-Poor Settings: Current and Future Implementation Challenges. Clin Infect Dis. 2016 Apr 15;62(8):1043-8. doi: 10.1093/cid/ciw001. Epub 2016 Jan 6. PMID 26743094
- [Background] Shafiee H, Wang S, Inci F, Toy M, Henrich TJ, Kuritzkes DR, Demirci U. Emerging technologies for point-of-care management of HIV infection. Annu Rev Med. 2015;66:387-405. doi: 10.1146/annurev-med-092112-143017. Epub 2014 Nov 12. PMID 25423597
- [Background] Ouattara EN, Robine M, Eholie SP, MacLean RL, Moh R, Losina E, Gabillard D, Paltiel AD, Danel C, Walensky RP, Anglaret X, Freedberg KA. Laboratory Monitoring of Antiretroviral Therapy for HIV Infection: Cost-Effectiveness and Budget Impact of Current and Novel Strategies. Clin Infect Dis. 2016 Jun 1;62(11):1454-1462. doi: 10.1093/cid/ciw117. Epub 2016 Mar 1. PMID 26936666
- [Background] Marseille E, Giganti MJ, Mwango A, Chisembele-Taylor A, Mulenga L, Over M, Kahn JG, Stringer JS. Taking ART to scale: determinants of the cost and cost-effectiveness of antiretroviral therapy in 45 clinical sites in Zambia. PLoS One. 2012;7(12):e51993. doi: 10.1371/journal.pone.0051993. Epub 2012 Dec 20. PMID 23284843